CLINICAL TRIAL: NCT01534832
Title: Assessment of a New Surgical Smoke Clearing Technology, "Innervision", in Laparoscopic Cholecystectomy
Brief Title: Assessment of a New Surgical Smoke Clearing Technology in Laparoscopic Cholecystectomy
Acronym: Innervision
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asalus Medical Instruments Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: AMIL/2011/INV01
Record Dates: First submitted 2012-02-10; First posted 2012-02-17 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Focus: Surgical Smoke During Laparoscopic Surgery
Keywords: surgical smoke; laparoscopic surgery; impaired vision
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Smoke clearance (Experimental): Smoke clearance device active
  Interventions: Device: Innervision Surgical Smoke Removal System

INTERVENTIONS:
Device: Innervision Surgical Smoke Removal System — Smoke removal by electrostatic precipitation

SUMMARY:
The study will examine the safety and performance of a new surgical smoke clearance system designed for use during laparoscopic surgery.

DETAILED DESCRIPTION:
The study will examine the safety and performance of a new surgical smoke clearance system which has been developed to maintain a visually clear operative field during laparoscopic surgery by using electrostatic precipitation to clear, from the surgical field, smoke and plume produced by energy based surgical instruments e.g. electrocautery, laser tissue ablation and ultrasonic scalpel tissue dissection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age
2. Undergoing elective laparoscopic cholecystectomy for documented symptomatic gallstone disease
3. Patient or authorised representative must be able to comprehend and sign the Informed Consent Form prior to enrolment in the study.

Exclusion Criteria:

1. <18 years of age
2. Pregnant or lactating females
3. Previous extensive abdominal surgery, which in the opinion of the Investigator presents a >5% risk of conversion to an open procedure being required
4. Current participation in another device or drug study
5. Unwilling or unable to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Maintenance of a clear visual field during surgery | 3m

CONTACTS AND LOCATIONS:
Overall Officials: Jared Torkington, MBBS MS FRCS, Principal Investigator — Cardiff and Vale UHB, Wales, UK
Locations (1):
- University Hospital Llandough, Cardiff, Wales, United Kingdom